CLINICAL TRIAL: NCT01290549
Title: An Open-Label, Multicenter, Phase I Trial of the Safety and Pharmacokinetics Of Escalating Doses of DCDS4501A in Patients With Relapsed or Refractory B-Cell Non-Hodgkins Lymphoma and Chronic Lymphocytic Leukemia and DCDS4501A in Combination With Rituximab in Patients With Relapsed or Refractory B-Cell Non-Hodgkins Lymphoma
Brief Title: A Study of Escalating Doses of Polatuzumab Vedotin in Participants With Relapsed or Refractory B-Cell Non-Hodgkins Lymphoma and Chronic Lymphocytic Leukemia and Polatuzumab Vedotin in Combination With Rituximab in Participants With Relapsed or Refractory B-Cell Non-Hodgkins Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCS4968g; GO01294 (Other: Hoffmann-La Roche); 2011-002330-39 (EudraCT Number)
Record Dates: First submitted 2011-02-03; First posted 2011-02-07 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Non-Hodgkins Lymphoma; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — polatuzumab vedotin; Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Polatuzumab Vedotin (Experimental): Polatuzumab vedotin will be administered by an IV infusion of escalating doses (starting dose of 0.1 mg/kg, potentially to be followed by 0.25 mg/kg, 0.5 mg/kg, 1.0 mg/kg, 2.0 mg/kg, and 4.0 mg/kg doses) every 3 weeks (q3w) (Day 1 of each 21 day cycle).
  Interventions: Drug: Polatuzumab Vedotin
- Polatuzumab Vedotin + Rituximab (Experimental): Polatuzumab vedotin will be administered by an IV infusion q3w (Day 1 of each 21 day cycle). Rituximab was administered by an IV infusion at 375 milligrams per square meter (mg/m^2) body surface area dose q3w.
  Interventions: Drug: Polatuzumab Vedotin; Drug: Rituximab

INTERVENTIONS:
Drug: Polatuzumab Vedotin — Participants will receive escalating intravenous dose of polatuzumab vedotin.
  Other Names: DCDS4501A
Drug: Rituximab — Rituximab will be administered by an IV infusion at 375 mg/m^2 body surface area dose q3w.
  Arms: Polatuzumab Vedotin + Rituximab

SUMMARY:
This is a Phase I, multicenter, open-label, dose-escalation study of polatuzumab vedotin administered as a single agent by intravenous (IV) infusion to participants with relapsed or refractory hematologic malignancies. In Phase Ib, participants will receive polatuzumab vedotin in combination with rituximab.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy of at least 12 weeks
* History of one of the following histologically-documented hematologic malignancy for which no effective standard therapy exists: indolent non Hodgkin's lymphoma (NHL), Grade 3b follicular lymphoma (FL), diffuse large B-cell lymphoma (DLBCL), mantle cell lymphoma (MCL), or chronic lymphocytic leukemia (CLL)
* All participants (NHL and B-cell chronic lymphocytic leukemia [B-CLL]) must have at least one bi-dimensionally measurable lesion
* For all men or women of childbearing potential (unless surgically sterile): use of adequate methods of contraception such as oral contraceptives, intrauterine device, or barrier method of contraception in conjunction with spermicidal jelly

Exclusion Criteria:

* Prior use of any monoclonal antibody or antibody-drug conjugate within 4 weeks before Cycle 1, Day 1
* Treatment with radiotherapy, any chemotherapeutic agent, or treatment with any other investigational anti-cancer agent within 2 weeks prior to Cycle 1, Day 1. Adverse events from any previous treatments must be resolved or stabilized prior to Cycle 1, Day 1, except for neuropathy
* Completion of autologous stem cell transplant within 100 days prior to Cycle 1, Day 1
* Prior allogeneic stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2011-03-22 (Actual); Primary Completion 2012-06-29 (Actual); Study Completion 2014-11-18 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Dose-Limiting Toxicities (DLTs) | Cycle 1 (Days 1-21)
Maximum Tolerated Dose | Cycle 1 (Days 1-21)
Proposed Phase II Dose of Polatuzumab Vedotin | Cycle 1 (Days 1-21)
Percentage of Participants With Adverse Events (AEs) | Baseline up to 646 Days

SECONDARY OUTCOMES:
Percentage of Paticipants with Anti Therapeutic Antibodies (ATAs) Against Polatuzumab Vedotin | Preinfusion (0 hour) on Day 1 of Cycles 1, 2, 4, and at the treatment completion/early termination visit (up to 646 days)
Progression Free Survival (PFS), as Assessed by Using Modified Response Criteria for Non-Hodgkin Lymphoma (NHL) or Chronic Lymphocytic Leukemia (CLL) | Baseline up to disease progression or death (Every 3 months while on study treatment from the initiation of therapy and 30 days after last dose of study drug [up to 44.5 months])
Percentage of Participants With Objective Response [Complete Response (CR) or Partial Response (PR)], as Assessed by Using Modified Response Criteria for NHL or CLL | Every 3 months while on study treatment from the initiation of therapy and 30 days after last dose of study drug (up to 44.5 months)
Duration of Response, as Assessed by Using Modified Response Criteria for NHL or CLL | Baseline up to disease progression or death (Every 3 months while on study treatment from the initiation of therapy and 30 days after last dose of study drug [up to 44.5 months])
Percentage of Participants with Best Overall Response (BOR), as Assessed by Using Modified Response Criteria for NHL or CLL | Baseline up to disease progression or death (Every 3 months while on study treatment from the initiation of therapy and 30 days after last dose of study drug [up to 44.5 months])
Area Under the Curve (AUC) from Time 0 to The Last Quantifiable Time Point (AUClast)-Polatuzumab Vedotin Monotherapy | Pre infusion (0 hour) and 0.5, 4 hours post infusion (duration of infusion: 90 minutes for first infusion and 30 minutes for subsequent infusions) on Cycle 1 Day 1; Cycle 1 Days 2, 4, 8, 11 and 15 (cycle length: 21 days)
AUC Extrapolating to Time of Infinity (AUCinf)-Polatuzumab Vedotin Monotherapy | Pre infusion (0 hour) and 0.5, 4 hours post infusion (duration of infusion: 90 minutes for first infusion and 30 minutes for subsequent infusions) on Cycle 1 Day 1; Cycle 1 Days 2, 4, 8, 11 and 15 (cycle length: 21 days)
Percentage of AUCinf (AUCextrap)-Polatuzumab Vedotin Monotherapy | Pre infusion (0 hour) and 0.5, 4 hours post infusion (duration of infusion: 90 minutes for first infusion and 30 minutes for subsequent infusions) on Cycle 1 Day 1; Cycle 1 Days 2, 4, 8, 11 and 15 (cycle length: 21 days)
Maximum Plasma Concentration (Cmax)-Polatuzumab Vedotin Monotherapy | Pre infusion (0 hour) and 0.5, 4 hours post infusion (duration of infusion: 90 minutes for first infusion and 30 minutes for subsequent infusions) on Cycle 1 Day 1; Cycle 1 Days 2, 4, 8, 11 and 15 (cycle length: 21 days)
Clearance-Polatuzumab Vedotin Monotherapy | Pre infusion (0 hour) and 0.5, 4 hours post infusion (duration of infusion: 90 minutes for first infusion and 30 minutes for subsequent infusions) on Cycle 1 Day 1; Cycle 1 Days 2, 4, 8, 11 and 15 (cycle length: 21 days)
Volume of Distribution at Steady State-Polatuzumab Vedotin Monotherapy | Pre infusion (0 hour) and 0.5, 4 hours post infusion (duration of infusion: 90 minutes for first infusion and 30 minutes for subsequent infusions) on Cycle 1 Day 1; Cycle 1 Days 2, 4, 8, 11 and 15 (cycle length: 21 days)
AUClast - Polatuzumab Vedotin Combined with Rituximab | Pre infusion (0 hour) and 0.5 hours post infusion (duration of infusion: 90 minutes for first infusion and 30 minutes for subsequent infusions) on Cycle 1 Day 1; Cycle 1 Days 2, 4, 8, 11 and 15 (cycle length: 21 days)
AUCinf-Polatuzumab Vedotin Combined with Rituximab | Pre infusion (0 hour) and 0.5 hours post infusion (duration of infusion: 90 minutes for first infusion and 30 minutes for subsequent infusions) on Cycle 1 Day 1; Cycle 1 Days 2, 4, 8, 11 and 15 (cycle length: 21 days)
AUCextrap-Polatuzumab Vedotin Combined with Rituximab | Pre infusion (0 hour) and 0.5 hours post infusion (duration of infusion: 90 minutes for first infusion and 30 minutes for subsequent infusions) on Cycle 1 Day 1; Cycle 1 Days 2, 4, 8, 11 and 15 (cycle length: 21 days)
Cmax-Polatuzumab Vedotin Combined with Rituximab | Pre infusion (0 hour) and 0.5 hours post infusion (duration of infusion: 90 minutes for first infusion and 30 minutes for subsequent infusions) on Cycle 1 Day 1; Cycle 1 Days 2, 4, 8, 11 and 15 (cycle length: 21 days)
Clearance-Polatuzumab Vedotin Combined with Rituximab | Pre infusion (0 hour) and 0.5 hours post infusion (duration of infusion: 90 minutes for first infusion and 30 minutes for subsequent infusions) on Cycle 1 Day 1; Cycle 1 Days 2, 4, 8, 11 and 15 (cycle length: 21 days)
Volume of Distribution at Steady State-Polatuzumab Vedotin Combined with Rituximab | Pre infusion (0 hour) and 0.5 hours post infusion (duration of infusion: 90 minutes for first infusion and 30 minutes for subsequent infusions) on Cycle 1 Day 1; Cycle 1 Days 2, 4, 8, 11 and 15 (cycle length: 21 days)
AUClast of Rituximab When Given in Combination With Polatuzumab Vedotin | Pre rituximab (0 hour) dose and 30 minutes post rituximab dose on Cycle 1 Day 1; Cycle 1 Days 4, 8, 15 (cycle length: 21 days)
AUCinf of Rituximab When Given in Combination With Polatuzumab Vedotin | Pre rituximab (0 hour) dose and 30 minutes post rituximab dose on Cycle 1 Day 1; Cycle 1 Days 4, 8, 15 (cycle length: 21 days)
AUCextrap of Rituximab When Given in Combination With Polatuzumab Vedotin | Pre rituximab (0 hour) dose and 30 minutes post rituximab dose on Cycle 1 Day 1; Cycle 1 Days 4, 8, 15 (cycle length: 21 days)
Cmax of Rituximab When Given in Combination With Polatuzumab Vedotin | Pre rituximab (0 hour) dose and 30 minutes post rituximab dose on Cycle 1 Day 1; Cycle 1 Days 4, 8, 15 (cycle length: 21 days)
Clearance of Rituximab When Given in Combination With Polatuzumab Vedotin | Pre rituximab (0 hour) dose and 30 minutes post rituximab dose on Cycle 1 Day 1; Cycle 1 Days 4, 8, 15 (cycle length: 21 days)
Volume of Distribution at Steady State-of Rituximab When Given in Combination With Polatuzumab Vedotin | Pre rituximab (0 hour) dose and 30 minutes post rituximab dose on Cycle 1 Day 1; Cycle 1 Days 4, 8, 15 (cycle length: 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Waye Chu, M.D., Study Director — Genentech, Inc.
Locations (16):
- United States (7):
  - Stanford Cancer Center, Stanford, California
  - Stanford Cancer Institute Pharmacy, Stanford, California
  - Florida Cancer Specialists; Sarasota, Sarasota, Florida
  - Roswell Park Cancer Inst., Buffalo, New York
  - Sarah Cannon Cancer Center, Germantown, Tennessee
  - M.D Anderson Cancer Center; Oncology, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Canada (3):
  - Cross Cancer Institute ; Dept of Medical Oncology, Edmonton, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - McGill University; Sir Mortimer B Davis Jewish General Hospital; Oncology, Montreal, Quebec
- France (5):
  - CHU Dijon - SCE Hemato, Dijon
  - Centre Hospitalier Regional Universitaire de Lille, Lille
  - CHU Lapeyronie, Hematologie, Montpellier
  - Centre Hospitalier Lyon Sud; Hematolgie, Pierre-Bénite
  - Centre Henri Becquerel; Hematologie, Rouen
- Academisch Medisch Centrum; Hematologie, Amsterdam, Netherlands

REFERENCES:
- [Derived] Shi R, Lu T, Ku G, Ding H, Saito T, Gibiansky L, Agarwal P, Li X, Jin JY, Girish S, Miles D, Li C, Lu D. Asian race and origin have no clinically meaningful effects on polatuzumab vedotin pharmacokinetics in patients with relapsed/refractory B-cell non-Hodgkin lymphoma. Cancer Chemother Pharmacol. 2020 Sep;86(3):347-359. doi: 10.1007/s00280-020-04119-8. Epub 2020 Aug 8. PMID 32770353
- [Derived] Lu T, Gibiansky L, Li X, Li C, Shi R, Agarwal P, Hirata J, Miles D, Chanu P, Girish S, Jin JY, Lu D. Exposure-safety and exposure-efficacy analyses of polatuzumab vedotin in patients with relapsed or refractory diffuse large B-cell lymphoma. Leuk Lymphoma. 2020 Dec;61(12):2905-2914. doi: 10.1080/10428194.2020.1795154. Epub 2020 Jul 24. PMID 32705923
- [Derived] Palanca-Wessels MC, Czuczman M, Salles G, Assouline S, Sehn LH, Flinn I, Patel MR, Sangha R, Hagenbeek A, Advani R, Tilly H, Casasnovas O, Press OW, Yalamanchili S, Kahn R, Dere RC, Lu D, Jones S, Jones C, Chu YW, Morschhauser F. Safety and activity of the anti-CD79B antibody-drug conjugate polatuzumab vedotin in relapsed or refractory B-cell non-Hodgkin lymphoma and chronic lymphocytic leukaemia: a phase 1 study. Lancet Oncol. 2015 Jun;16(6):704-15. doi: 10.1016/S1470-2045(15)70128-2. Epub 2015 Apr 27. PMID 25925619
- See also: Link to the publication — https://www.ncbi.nlm.nih.gov/pubmed/25925619?dopt=Abstract